CLINICAL TRIAL: NCT00005699
Title: Improving Hypertension Control in the Inner City
Status: Completed | Type: Observational
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Sponsor
Other Study IDs: 4278
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-02-11 (Estimated); Status verified 2016-02

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Hypertension
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Hypertensive: described as hypertensive according to AHA guidelines at time of trial
- Controls: described as non-hypertensive according to AHA guidelines at time of trial

SUMMARY:
To conduct a community based education program using existing resources to improve hypertension control in the inner city through multiple interventions.

DETAILED DESCRIPTION:
BACKGROUND:

The study was in response to a demonstration and education initiative, "Improving Hypertensive Care for Inner City Minorities", which was reviewed and approved by the Clinical Applications and Prevention Advisory Committee in April 1992 and by the National Heart, Lung, and Blood Advisory Council in May 1992. The Request for Applications was released in October 1992.

DESIGN NARRATIVE:

The program consisted of a community wide education program, an intensive intervention directed toward individuals with hypertension, and an intervention for health care providers. The program was developed by a coalition of community organizations. In the community wide educational intervention, a baseline household survey was used to identify barriers to hypertension control in the community. This information was used in planning the intervention strategies, targeting the educational efforts, and developing the educational messages. Existing community organizations (churches, local media, neighborhood organizations, etc) were used to implement educational efforts over a three year period. Program success was evaluated by comparing findings on a follow-up household survey with those at baseline. Level of blood pressure control was the primary outcome measure. For the intensive educational program for hypertensives, the investigators developed a hypertension registry of individuals with high blood pressure who were identified from a number of community sources. All individuals on the registry receive educational material through the mail. Individuals with uncontrolled hypertension were randomized to receive the usual mailed educational materials or a more intensive personalized 12 month intervention using lay health advisors.

In the evaluation, the investigators compared blood pressure control morbidity and mortality between these two intervention arms of the registry. The innovative educational approach to health care providers utilized the existing community-based Area Health Education Center (AHEC) network to communicate community-determined hypertension control needs and community-determined hypertension control strategies to health care providers and students. The research was designed to elucidate community factors in the inner city that dictated strategies necessary for success in a variety inner city environments. Specifically, the investigators examined the effect of community size and level of community stress (as indicated by poverty, crime, etc.) on program development and outcome. To do this, they implemented the program in one city-wide community (Milwaukee) and in three well defined, homogeneous inner city neighborhoods of Chicago which had differing levels of community stress indicators. They evaluated the effect of size and community stress levels on the program strategies and successes.

ELIGIBILITY:
No eligibility criteria

Ages: 18 Years to 100 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: African-Americans with or without hypertension
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Actual)
Dates: Start 1993-09; Primary Completion 2005-02 (Actual); Study Completion 2005-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jane Kotchen, Principal Investigator — Medical College of Wisconsin

IPD SHARING:
Plan to Share IPD: Undecided
to be published

REFERENCES:
- [Background] Kotchen JM, Shakoor-Abdulllah B, Walker W, Peters B, Kotchen TA. Planning for a community-based hypertension control program in the inner city. J Hum Hypertens. 1996 Sep;10 Suppl 3:S9-13. PMID 8872817
- [Background] Kotchen JM, Shakoor-Abdullah B, Walker WE, Chelius TH, Hoffmann RG, Kotchen TA. Hypertension control and access to medical care in the inner city. Am J Public Health. 1998 Nov;88(11):1696-9. doi: 10.2105/ajph.88.11.1696. PMID 9807539
- [Background] Shakoor-Abdullah B, Kotchen JM, Walker WE, Chelius TH, Hoffmann RG. Incorporating socio-economic and risk factor diversity into the development of an African-American community blood pressure control program. Ethn Dis. 1997 Autumn;7(3):175-83. PMID 9467699